# **Informed Consent**

Title:

Comparative Analysis of Different Physiotherapy Interventions on Anterior Pelvic Tilt in Subjects with Non-Specific Low Back Pain: A Randomized Controlled Trial

## Appendix A

## **Informed consent Form**

- 1. **Title of study**: Comparative Analysis of different physiotherapy Interventions on Anterior Pelvic Tilt in Subjects with Non-Specific Low Back Pain: A Randomized Controlled Trial
- 2. Name of investigator: Mahtab Ahmad Mukhtar Patafi
- 3. Name of Institution: Lincoln University, Malaysia

## 4. Introduction:

You should be aware of the reasons behind the research and the scope of it as well. Before deciding whether you are ready to join, kindly review and give great thought to this material. Enquire about the study team whether something seems unclear or whether you would want more information. You must complete this informed consent form after you are sufficiently convinced you understand this study and you want to take part.

You entered this research voluntarily. Should you not want to participate in this study, you are not required to. You might simply refuse to respond to any questions you wish not to address. Should you volunteer for this study, you are free to withdraw at any point. Should you withdraw, the information gathered from you up to that point will still be used for the study. Your non-participation or withdrawal has no bearing on any medical or health benefit for which you are otherwise entitled.

The Research and Ethics Committee of Licoln University College, Malaysia as well as National Hospital, Bahawalpur will allow this study.

## 5. What is the Objective of the study?

The purpose of this study is to assess and compare the effects of different physiotherapy modalities, including dry needling, manual mobilization and soft tissue release, trigger point therapy, stretching, cupping therapy, and electrotherapy, on the craniovertebral angle in individuals diagnosed with myofascial pain syndrome (MPS) and radiculopathy. This research is necessary to improve the understanding of parents of children with Autism.

This research will be conducted for a duration of 06 months (16/11/2024 till 15/07/2025). The expected number of participants is 100 individuals.

## 6. What are my responsibilities when taking part in this study?

It will take roughly ten minutes of your time to honestly and totally answer all the questions posed by the research crew. The study team will also access your medical records for the following information.

- Previous medical history
- Previous surgical history
- Previous history of trauma
- History of any chronic condition

You will be given a survey form to be answered. This form contains eight sections which will enquire about your health status and quality of life.

## 7. What are the potential risks and side effects of being in this study?

Participation to this study will not affect your treatment, and the risk is minimal. You are free to decline to answer any of the questions that you feel uncomfortable with.

## 8. What are the benefits of being in this study?

There may or may not be any benefits to you. Information obtained from this study will help to decide the treatment options for myofascial pain syndrome and radiculopathy.

## 9. Who is funding the research?

This study is sponsored by none other than the researcher himself. You will not be paid for participating in this study.

## 10. Will my medical information be kept private?

11. In line with relevant laws and/or guidelines, all the information you gather for this study will be stored and managed in a private manner. Your identity won't be revealed without your stated permission when publishing or presenting the study findings. Those engaged in this research, qualified auditors and monitors, government or regulatory bodies, could review the study data, when relevant and required.

## 12. Who should I call if I have questions?

If you have any questions about the study or if you think you have a study related injury and you want information about this study, please contact the study doctor, Mahtab Ahmad Mukhtar Patafi at telephone number +92-301-7766019.

#### INFORMED CONSENT FORM

Title of Study: Comparative Analysis of Physiotherapy Treatments on Craniovertebral Angle in Individuals with Myofascial Pain Syndrome and Radiculopathy: A Randomized Controlled Trial

By signing below, I confirm the following:

- I have been given oral and written information for the above study and have read and understood the information given.
- I have had sufficient time to consider participation in the study and have had the opportunity to ask questions, and all my questions have been answered satisfactorily.
- I am aware that my involvement is voluntary and that I can at any moment freely withdraw from the study without stating a reason; this will not in any way influence my future treatment. At right moment, I am not participating in any other research project. Knowing the risks and rewards, I willingly provide my informed permission to take part under the specified terms. I am aware that I must do as advised by the study doctor—investigator—about my involvement in the study.
- I am aware that direct access to my medical record is granted to study staff, qualified monitors and auditors, sponsors or associates, government or regulatory bodies, therefore ensuring proper operation of the study and accurate data recording. Every personal information will be handled as strictly confidentially.
- I will receive a copy of this subject information/informed consent form signed and dated to bring home.
- I agree/disagree for my family doctor to be informed of my participation in this study.

## **Subject:**

| Signature: | I/C number: |
|-------------------------------------------|-------------|
| Name: | Date: |
| Investigator conducting informed consent: | |
| Signature: | I/C number: |
| Name: | Date: |